CLINICAL TRIAL: NCT07119385
Title: Quasi-experimental Pre-post Study Assessing the Impact of Non-pharmacological Interventions Based on Nursing Care and of an Educational Programme for Delirium Prevention in Older Adults With Cognitive Frailty During Hospitalization
Brief Title: Non-pharmacological Measures for the Prevention of Delirium in Frail Hospitalized Adults. Nursing Care (PREDELENF)
Acronym: PREDELENF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PI-23-105
Record Dates: First submitted 2025-06-27; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Delirium in Old Age
Keywords: Prevention; Delirium; Frailty; Multicomponent intervention
MeSH Terms: conditions — Delirium; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (usual medical care) (Other): The usual care will be provided according to the center's protocols.
  Interventions: Other: Usual care
- Intervention (PREDELENF Multicomponent Intervention) (Experimental): A multicomponent intervention designed for the prevention of delirium in frail patients.Include different actions (see variables)
  Interventions: Other: Multicomponent non-pharmacological interventions

INTERVENTIONS:
Other: Multicomponent non-pharmacological interventions — Multicomponent non-pharmacological interventions to prevent delirium in frail patients
  Arms: Intervention (PREDELENF Multicomponent Intervention)
Other: Usual care — Usual care
  Arms: No intervention (usual medical care)

SUMMARY:
Background: Delirium is one of the most frequent, relevant, and increasing geriatric syndromes in hospitalized older adults. It is an indicator of poor prognosis, and its incidence increases with aging. It is a highly prevalent problem (between 10-56% of hospitalized elderly), underdiagnosed (32-66% undetected), with severe consequences and potentially preventable (between 30-40%). It is considered a priority health objective, as it is an indicator of elderly patient safety and an indicator of healthcare quality.

Objective: The objective of this study is to analyze whether a multicomponent nursing-led intervention reduces the incidence of delirium in frail older patients hospitalized in a medical unit.

Design: Pre-post quasi-experimental analytical study. Study setting: The study will be conducted in a polyvalent hospitalization unit at the Germans Trias i Pujol University Hospital during the 2023-2025 period.

Patients: A total of 158 patients will be needed, i.e., 79 for each group. Sampling: Consecutive intentional sampling based on inclusion and exclusion criteria.

Variables: Sociodemographic variables, delirium risk factors, daily presence of delirium using the CAM scale, and hospital stay duration, among others, will be collected.

Procedure: Patients will be selected upon admission, and the presence of delirium will be assessed daily using the CAM scale, with results recorded. Nursing staff will be trained on non-pharmacological measures for delirium prevention and a specific care plan. Subsequently, the second group of patients will receive these specific interventions, and the presence of delirium will be assessed daily using the CAM scale, with results recorded.

Data analysis: Descriptive and inferential analysis using the PSPP statistical package version 22. A significance level of 5% will be applied.

DETAILED DESCRIPTION:
A pre-post quasi-experimental study will be conducted with a control group and an intervention group. Consecutive sampling will be performed purposively, using inclusion and exclusion criteria. A total of 158 patients are required, i.e., 79 per group. Granmo software was used to calculate the sample. An alpha risk of 0.05 was assumed, with a two-sided contrast and a beta risk of 0.2. The allocation ratio will be 1, and a 10% loss to follow-up rate and a 20% reduction in the incidence of delirium have been estimated.

Participants Patients over 70 years of age admitted to the HGTIP study units for conditions requiring hospitalization and who meet the established criteria. The inclusion and exclusion criteria for selecting participants for this study are shown in Table 1.

Recruitment of participants Candidates for the study will be identified daily by a member of the research team, who will check the computerized devices used to detect new admissions to the study unit. Those who meet the inclusion criteria will be invited to participate. The study will be explained to them, including their family members. If they agree, they will be provided with an informed consent form, which they will sign.

All patients admitted to the study unit who meet the established criteria will be included in the sample, until the required sample size is reached, estimated at approximately six months for the control group and another six months for the intervention group.

Intervention The study will be conducted in the multipurpose hospitalization unit of the Germans Trias i Pujol University Hospital (HUGTIP) during the period 2024-2025.

A. First, data will be collected to analyze the incidence of delirium in the unit prior to the intervention (baseline data/usual care).

B. The work to be performed will be communicated to the nursing and medical specialty teams of the multipurpose hospitalization unit and will be presented as an intervention to improve the quality of care.

C. A 1-hour in-person training program will be provided for each work shift (morning, afternoon, evening 1, and evening 2) to all professionals in the intervention unit.

D. Implementation of the multicomponent care plan specific to the prevention of delirium. (Annex 3).

E. The impact of training on clinical outcomes in the intervention unit will be analyzed.

F. Finally, the incidence of delirium will be analyzed, along with the specific care plan and training for professionals in preventing the syndrome.

Elements of the investigation A multicomponent care plan has been designed, comprising 12 intervention areas based on the main risk factors for delirium. For each area, different activities are proposed, as shown in Table 2. The intervention also includes a series of structural and scheduling modifications in the study unit, as specified in Table 3.

Furthermore, the training program that will be provided to all professionals in the intervention unit is based on strategies recommended by the Spanish Society of Geriatrics and Gerontology (SEGG) for the prevention of delirium.

The training will include the definition of delirium, symptoms of delirium that will help us recognize it early, its presentation (hyperactivity, hypoactivity, and mixed forms), training in the detection of delirium using the CAM scale, possible causes, predisposing and precipitating factors, the evolution of delirium once it has developed, prevention strategies, non-pharmacological measures, and the use of medications.

Implementation of the intervention The control group's data collection period will last approximately six months, or until the required sample size is reached. The unit's professionals will then be informed about the work to be performed, and their knowledge of the topic will be analyzed through a survey. The training program will then be delivered, and the care plan, along with any structural and scheduling modifications, will be implemented. Participants will be asked to complete the knowledge survey again to evaluate the training's impact. Finally, data will be collected from the intervention group for approximately another six months, or until the full sample size is reached.

Data collection Data collection will be conducted by the same professional from the research team within the first 24 to 48 hours of admission, based on medical records, nursing records, and information obtained directly from the patient and support staff.

Upon admission, sociodemographic data will be collected (age, sex, origin: home, intermediate care, residence, admission diagnosis and global status (Charlson, Pfeiffer, Barthel, Rockwood/CFS, PCC, ECA and presence of geriatric syndromes such as dysphagia, incontinence, falls, and other factors predisposing to delirium such as cognitive impairment, depression, pain, sensory disturbances, nutritional status, dehydration, delirium in previous admissions, psychoactive medication).

Daily data collection during admission includes the following variables: presence of delirium using the CAM scale, follow-up, correction of sensory disturbances, cognitive stimulation, mobilization, hydration and nutrition, psychoactive medications, and nighttime rest.

The variables to be collected for discharge are: days of admission, presence of delirium, days of duration of delirium, Pfeiffer, Barthel, destination: home, intermediate care, residence, psychoactive medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients >70 years old
* Conscious mental state. And one of the two criteria described below:
* Pfeiffer score on admission between 3-7 errors, according to the nursing assessment within the first 24 hours of admission to the ward, suggesting possible mild-moderate cognitive impairment.
* Any degree of diagnosed dementia, except GDS7.

Exclusion Criteria:

* Patients unable to communicate, with established aphasia, or with psychiatric illness.
* Patients with a language barrier.
* Patients transferred from other units.
* Terminal situation under palliative treatment.
* Patients who do not consent to participate

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 158 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Presence of Delirium | From baseline (day 1) until day 12 (expected date of hospital discharge or death from any cause)
  Assessment of the presence of delirium will be performed by trained personnel using the Confusion Assessment Method (CAM). The CAM consists of four items, and a positive CAM (indicating the presence of delirium) is defined as the presence of both of the first two items (1 and 2) and at least one of the last two items (3 or 4).

SECONDARY OUTCOMES:
Sociodemographic Variables | Baseline
  Gender, age, and place of origin (home, nursing home)
Current illness/geriatric assessment upon admission. Assess cognition using the Pfeiffer Questionnaire | Baseline
  The Pfeiffer Questionnaire is a screening tool used to detect cognitive impairment. It consists of 10 items, and a score of three or more may indicate cognitive impairment. Higher scores are associated with a greater likelihood of cognitive decline
Current illness/geriatric assessment upon admission. Diagnosis of Dementia | Baseline
  Review the patient's medical record for a diagnosis of dementia prior to admission
Current illness/geriatric assessment upon admission. Degree of frailty | Baseline
  The Rockwood Clinical Frailty Scale (CFS) is a scoring tool that assesses frailty using a 9-point scale. The higher the score, the greater the patient's level of frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Moreno, RN,MSC,PhDc, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobar E, Alvarez E. Delirium en el adulto mayor hospitalizado. RMCLC. 2020;
- [Background] Chavez-Delgado ME, Virgen-Enciso M, Perez-Guzman J, Celis-de-la-Rosa A, Castro-Castaneda S. [Detection of delirium in hospitalized elderly patients using the confusion assessment method]. Rev Med Inst Mex Seguro Soc. 2007 Jul-Aug;45(4):321-8. Spanish. PMID 17949569
- [Background] Cano G. Contribuciones al estudio de factores de riesgo y mortalidad del delirium y fragilidad en adultos mayores hospitalizados. Bilbao. 2022.
- [Background] Fernandez Mª, Faus M. Medidas no farmacológicas para la prevención del delirium en pacientes ingresados en Unidades de Cuidados Intensivos. THERAPEÍA. 2021;14: 113-40.
- [Background] Gonzalez B, Marín JM, Gutierrez V, Velilla N. Protocolo diagnóstico y manejo del delirium en el anciano. Protocolos. 2018;12(62): 3670-4.
- [Background] Carrasco G M, Villarroel D L, Calderon P J, Martinez F G, Andrade A M, Gonzalez T M. [Development and validation of a clinical predictive model for delirium in hospitalized older people]. Rev Med Chil. 2014 Jul;142(7):826-32. doi: 10.4067/S0034-98872014000700002. Spanish. PMID 25378001
- [Background] Restrepo D, Duque M, Montoya L, Berrouet MC, Rojas M, Lopera G, Giraldo K. Risk Factors and Hospital Mortality in Surgical and Non-surgical Patients with Delirium. Rev Colomb Psiquiatr (Engl Ed). 2018 Jul-Sep;47(3):148-154. doi: 10.1016/j.rcp.2017.03.001. Epub 2017 Apr 21. English, Spanish. PMID 30017037
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Bellelli G, Brathwaite JS, Mazzola P. Delirium: A Marker of Vulnerability in Older People. Front Aging Neurosci. 2021 Apr 30;13:626127. doi: 10.3389/fnagi.2021.626127. eCollection 2021. PMID 33994990
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Carrasco M, Accatino-Scagliotti L, Calderon J, Villarroel L, Marin PP, Gonzalez M. [Delirium in older medical inpatients: a one year follow up study]. Rev Med Chil. 2012 Jul;140(7):847-52. doi: 10.4067/S0034-98872012000700003. Spanish. PMID 23282695
- [Background] Formiga F, San Jose A, Lopez-Soto A, Ruiz D, Urrutia A, Duaso E. [Prevalence of delirium in patients admitted because of medical conditions]. Med Clin (Barc). 2007 Oct 27;129(15):571-3. doi: 10.1157/13111707. Spanish. PMID 17988613
- [Background] Pão-Mole M, Dourado RM, Pontífice P. Delirium: intervenciones de enfermería en el adulto hospitalizado - una revisión bibliográfica. Enferm glob. 2018;17(52): 640-88.
- [Background] Perello Campaner C. [Delirium risk assessment in elderly hospitalized patients]. Rev Esp Geriatr Gerontol. 2010 Sep-Oct;45(5):285-90. doi: 10.1016/j.regg.2010.03.011. Epub 2010 Aug 8. Spanish. PMID 20696498
- [Background] Avendaño A. Ensayo clínico piloto de una intervención multicomponente de enfermería para reducir el delirium en ancianos hospitalizados. (MID-Nurse-P). Albacete. 2019
- [Background] Ramón JL, Gallardo M. Delirium o síndrome confusional agudo. AMF. 2015;11(9): 516-23
- [Background] Giraldo CC, Pérez JM, Sánchez DM. Terapia Física Temprana para la Prevención del Delirio en la Unidad de Cuidados Intensivos. Arch de Medicina. 2021;17(5): 1
- [Background] Carrera C, Romero FJ, González A. Revisión de la utilidad y fiabilidad de la Confusion Assessment Method en atención especializada y primaria, 2013. Av Enferm. 2015;33(2): 261-70.
- [Background] Miranda F, Gonzalez F, Plana MN, Zamora J, Quinn TJ, Seron P. Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) for the diagnosis of delirium in adults in critical care settings. Cochrane Database Syst Rev. 2023 Nov 21;11(11):CD013126. doi: 10.1002/14651858.CD013126.pub2. PMID 37987526
- [Background] Palihnich K, Gallagher, J, Inouye SK, Marcantonio ER. The 3D CAM Training Manual for Research. V4.1. 2016; Boston: Hospital Elder Life Program.
- [Background] Avendano-Cespedes A, Garcia-Cantos N, Gonzalez-Teruel Mdel M, Martinez-Garcia M, Villarreal-Bocanegra E, Oliver-Carbonell JL, Abizanda P. Pilot study of a preventive multicomponent nurse intervention to reduce the incidence and severity of delirium in hospitalized older adults: MID-Nurse-P. Maturitas. 2016 Apr;86:86-94. doi: 10.1016/j.maturitas.2016.02.002. Epub 2016 Feb 8. PMID 26921934
- [Background] Recasens-López M, Villamor-Ordozgoiti A, Sanz-Díez M, Sánchez-Morillo M, Serna-Landete R, Asensio-Rubio Y. Eficacia de un plan de cuidados de enfermería específico para el paciente con delirio. Rev Cubana Enfermer. 2019;35(1).
- [Background] Hshieh TT, Yang T, Gartaganis SL, Yue J, Inouye SK. Hospital Elder Life Program: Systematic Review and Meta-analysis of Effectiveness. Am J Geriatr Psychiatry. 2018 Oct;26(10):1015-1033. doi: 10.1016/j.jagp.2018.06.007. Epub 2018 Jun 26. PMID 30076080
- [Background] Sánchez E. Prevención del delirium en el paciente anciano: diseño y evaluación de una intervención no farmacológica en el ámbito hospitalario. Universidad Complutense de Madrid. 2015.
- [Background] Carrera C. Rol de enfermería en la prevención del delirium en ancianos hospitalizados con fractura de cadera: Recomendaciones generales. Enferm glob. 2012;11(27): 356-78.